CLINICAL TRIAL: NCT04922736
Title: Patient Reported Outcomes With UVA-1 Therapy for Treatment of Sclerosing Skin Diseases
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Christopher B Hansen, Assistant Professor, Dermatology, Principal Investigator, University of Utah
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB_00142027
Record Dates: First submitted 2021-06-08; First posted 2021-06-11 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Scleroderma, Systemic; Morphea; Graft Vs Host Disease
MeSH Terms: conditions — Scleroderma, Systemic; Scleroderma, Localized; Graft vs Host Disease

STUDY DESIGN:
Intervention Model Description: Single Group, open label,
Masking Description: No masking
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: UVA-1 Phototherapy — All patients will receive UVA-1 Phototherapy treatments

SUMMARY:
The purpose of this study is to assess the degree of improvement seen patient reported outcomes after 30 sessions of UVA-1 therapy in treating systemic scleroderma, morphea, and sclerodermatous Graft-Versus-Host Disease.

While patients have verbally reported improvement of their sclerosing skin disease with UVA-1, patient reported outcomes have not been rigorously studied. In sclerosing skin diseases where clinical change is difficult to measure, patient reported outcomes may offer a better way to study the impact of treatments like UVA-1.

This will be a non-blinded, non-randomized prospective trial using UVA-1 phototherapy in patients with established sclerosing skin disease. Patients will report the severity of their condition using multiple patient reported outcomes and will also be analyzed using multiple clinical investigator assessments at the beginning and end of 30 treatment sessions.

DETAILED DESCRIPTION:
Ultraviolet (UV) therapy has been used in dermatology for decades. UVA-1 phototherapy uses the longest wavelengths in the UV spectrum from 340-400 nm. It can penetrate the skin deeper than other types of phototherapy and target different cell types including fibroblasts. In sclerosing skin conditions UVA-1 appears to be superior to other forms of UV therapy. Medium-to-high dose UVA-1 also appears to be superior to low dose UVA-1 for sclerosing conditions.

Sclerosing skin diseases treated with UVA-1 include systemic sclerosis (SSc), morphea and sclerodermatous graft vs. host disease (GVHD). These are immune-mediated conditions that lead to skin fibrosis and may be associated with significant morbidity. These conditions share some common features including fibrotic skin changes that may have an active inflammatory stage followed by induration and scarring. Due to the depth of skin involvement, clinical assessment of the degree of active inflammation and depth of involvement is often challenging.

SSc, also called scleroderma, is a rare chronic autoimmune disease that can have a wide range of cutaneous, joint, and internal organ involvement. In the skin, SSc is characterized by enhanced fibroblast activity leading to hypertrophic dermal collagen that results in thickened, less flexible skin. SSc is often divided into two types based on extent of skin involvement: diffuse SSc and limited SSc. Morphea has similar cutaneous changes to SSc but lacks the internal organ involvement. Some of the common subtypes of morphea include circumscribed, linear, and generalized. Sclerodermatous GVHD, a complication of allogenic bone marrow or peripheral blood stem cell transplants, results in fibrotic skin changes that can be widespread and cause morbidity.

Multiple studies report skin improvement in these conditions using UVA-1. This improvement likely involves both dampening inflammation and reducing fibrosis. However, these studies generally lack validated clinical outcome measures. Development of these outcome measures has been slowed by the lack of tools to adequately assess change. Physician assessment, clinical scores, medical imaging, and tools such as a durometer have all been used to attempt to objectively measure changes with therapy over time, but all have limitations.

Patient reported outcomes (PROs) have attracted significant attention in clinical research in the past decade and are required by the FDA for clinical trials. These instruments refer to health outcomes reported directly by the patient who experienced the intervention. Established and validated PRO measures exist and have been used to evaluate multiple medical treatments. While patients have verbally reported improvement of their sclerosing skin disease with UVA-1, PROs have not been rigorously studied. In sclerosing skin diseases where clinical change is difficult to measure, PROs may offer a better way to study the impact of treatments like UVA-1.

Purpose and Objectives:

1. Primary objective: To assess the degree of improvement seen in the Health Assessment Questionnaire Disability Index (HAQ-DI) after 30 sessions of UVA-1 therapy in treating SSc, morphea, and sclerodermatous GVHD.
2. Secondary objectives: After 30 sessions of UVA-1 therapy:

   1. Assess changes in the Hand Mobility in Scleroderma (HAMIS) score in patients with hand involvement.
   2. Assess changes in the Localized Scleroderma Assessment Tool (LoSCAT) score in morphea patients.
   3. Assess changes in the Modified Rodnan Skin Score (mRSS) in SSc patients.
   4. Assess changes in the National Institutes of Health (NIH) Likert scale score in GVHD patients.
   5. Assess changes in durometer scores in all patients.
   6. Assess changes in PROs
   7. Compare changes in HAQ-DI scores to changes in LoSCAT, mRSS, NIH Likert scale, durometer, and HAMIS scores, as indicated

Study Design:

This will be a non-blinded, non-randomized prospective trial using UVA-1 phototherapy in patients with established sclerosing skin disease. Patients will report the severity of their condition using multiple PROs and will also be analyzed using multiple clinical investigator assessments at the beginning and end of 30 treatment sessions. In order to more accurately assess the outcome of UVA-1 therapy for each of the three different diseases, patients will be evaluated at the beginning and the end of the study using clinical scoring methods specific to each of the three diseases. Morphea patients will be assessed using LoSCAT, a reliable tool that captures disease activity and damage by assessing skin thickness, erythema, and new lesions/lesion extension. SSc disease activity and severity is more accurately assessed by measuring skin thickness. We will use a specific tool for SSc patients called the modified Rodnan's Skin Score (mRSS), which measures skin thickness on 17 different body areas. Disease activity for GVHD patients differs from morphea and SSc in that this GVHD affects multiple internal organ systems in addition to the skin; thus, a standardized measure is lacking for assessing skin-specific GVHD. Measures such as the MRSS and LoSCAT are also not recommended in clinical trials given these tests' inability to adequately assess the range of sclerotic changes seen in GVHD. Responses to the 2014 NIH criteria for assessing organ involvement in GVHD suggest assessing GVHD sclerotic skin disease activity with a clinician-reported 11-point scale of disease severity. We will therefore use this method and limit the assessment of GVHD patients to a single clinician to eliminate interrater variability. Additional clinical assessments for all patients will include durometry to assess skin hardness and the HAMIS test to assess hand function.

This is a prospective, single arm, clinical trial of UVA-1 therapy for multiple sclerosing skin conditions over 30 treatment sessions. The study will be performed at the University of Utah Dermatology Midvalley Clinic space where the UVA-1 light box is located. Personnel involved in the study will include the PI, the co-investigators, and the study coordinators.

At least 18 participants are needed to account for a 25% drop-out rate, although we plan to recruit 30 in total given the study funding available to meet the costs of all participants' treatments.

ELIGIBILITY:
Inclusion criteria:

* Must be able to understand and provide written informed consent
* Must have a diagnosis of systemic scleroderma with cutaneous sclerosis, morphea, or sclerodermatous Graft vs. host disease based on the presence of characteristic clinical findings
* Age of at least 18-years-old
* Ability to engage in 30 UVA-1 treatments in a maximum of 100 days.

Exclusion criteria:

* Inability to complete study visits
* UV light therapy in the 4 weeks prior to entering the study
* Commercial tanning in the 4 weeks prior to entering the study
* Current pregnancy or planned pregnancy during the study period
* History of intolerance to ultraviolet light
* Any other condition that will disqualify the patient from the study in the opinion of the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-06-07 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Evaluate change in the Health Assessment Questionnaire Disability Index (HAQ-DI) after 30 sessions of UVA-1 therapy in treating systemic Scleroderma, morphea, and sclerodermatous graft vs. host disease. | 100 days
  The Health Assessment Questionnaire Disability Index (HAQ-DI) is a validated patient self-administered tool used to assess changes in disease activity, especially the skin involvement in SSc (Steen, 1997). The questionnaire consists of 20 items in eight domains related to measuring the difficulty of performing activities of daily living, with each question rated on a scale of 0-3; 0 indicates "without difficulty" and 3 indicates "unable to do" (Allanore 2020).

SECONDARY OUTCOMES:
Assess changes in the Hand Mobility in Scleroderma (HAMIS) score in patients with hand involvement after 30 sessions of UVA-1 therapy. | 100 days
  HAMIS is a hand function test developed for adults with SSc and consists of 9 items designed to measure all movements assessed in an ordinary range of motion (ROM)-measured hand test. Specific items test finger flexion and extension, thumb abduction, pincer grip, finger abduction/swelling, dorsal extension and volar extension of the wrist, and pronation and supination. Each item is graded on a 0-3 scale, where 0 corresponds to normal function and 3 denotes that the individual is unable to perform the item. Each hand is assessed separately. The minimum score for HAMIS is 0, representing normal hand function. The maximum score is 27, representing a high degree of dysfunction (Sandqvist, 2000).
Assess changes in the Localized Scleroderma Assessment Tool (LoSCAT) score in morphea patients after 30 sessions of UVA-1 therapy. | 100 days
  The Localized Scleroderma Assessment Tool (LoSCAT) is a reliable tool to capture morphea disease activity and damage by assessing skin thickness, erythema, and new lesions/lesion extension. This tool assesses 18 different body locations using a 0-3 point scale, where 0 indicates no disability and 3 indicates complete disability (Skrzypek-Salamon, 2018). The score is calculated by adding the scores at each site to equal a total score ranging from 0 (normal) to 54 (severe disease).
Assess changes in the Modified Rodnan Skin Score (mRSS) in systemic scleroderma patients after 30 sessions of UVA-1 therapy. | 100 days
  The physician assessment on skin thickness based on the modified Rodnan skin score (mRSS) is a standard outcome measure for skin disease in systemic sclerosis. The score is calculated by evaluating the skin thickness at 17 different body sites. Each site is graded from 0 to 3, with 0 representing normal skin and 3 representing severe skin thickness. The score is calculated by adding the scores at each site to arrive at a total score ranging from 0 (normal) to 51 (severe disease) (Khanna, 2017).
Assess changes in the National Institutes of Health (NIH) Likert scale score in GVHD patients after 30 sessions of UVA-1 therapy. | 100 days
  The NIH severity score was created for assessing organ involvement in GVHD. Sclerotic skin disease is rated on an 11-point (0- to 10-point scale), clinician-reported assessment of disease severity (Lee, 2015). We will use this method and limit the assessment of patients with GVHD to a single clinician to eliminate interrater variability.
Assess changes in durometer scores in all patients after 30 sessions of UVA-1 therapy. | 100 days
  A Durometer is an instrument used to test the hardness of various materials. It has been used in scleroderma to compare the hardness of affected skin vs. normal skin. We will take an average of three durometry measurements at each of the involved sites.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher B. Hansen, M.D., Principal Investigator — University of Utah MidValley Dermatology
Locations (1):
- University of Utah Dermatology, Murray, Utah, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kreuter A, Hyun J, Stucker M, Sommer A, Altmeyer P, Gambichler T. A randomized controlled study of low-dose UVA1, medium-dose UVA1, and narrowband UVB phototherapy in the treatment of localized scleroderma. J Am Acad Dermatol. 2006 Mar;54(3):440-7. doi: 10.1016/j.jaad.2005.11.1063. Epub 2006 Jan 30. PMID 16488295
- [Background] Hassani J, Feldman SR. Phototherapy in Scleroderma. Dermatol Ther (Heidelb). 2016 Dec;6(4):519-553. doi: 10.1007/s13555-016-0136-3. Epub 2016 Aug 12. PMID 27519050
- [Background] Poole JL, Steen VD. The use of the Health Assessment Questionnaire (HAQ) to determine physical disability in systemic sclerosis. Arthritis Care Res. 1991 Mar;4(1):27-31. doi: 10.1002/art.1790040106. PMID 11188583
- [Background] Filippetti M, Cazzoletti L, Zamboni F, Ferrari P, Caimmi C, Smania N, Tardivo S, Ferrari M. Effect of a tailored home-based exercise program in patients with systemic sclerosis: A randomized controlled trial. Scand J Med Sci Sports. 2020 Sep;30(9):1675-1684. doi: 10.1111/sms.13702. Epub 2020 May 11. PMID 32350931
- [Background] Khanna D, Spino C, Johnson S, Chung L, Whitfield ML, Denton CP, Berrocal V, Franks J, Mehta B, Molitor J, Steen VD, Lafyatis R, Simms RW, Gill A, Kafaja S, Frech TM, Hsu V, Domsic RT, Pope JE, Gordon JK, Mayes MD, Schiopu E, Young A, Sandorfi N, Park J, Hant FN, Bernstein EJ, Chatterjee S, Castelino FV, Ajam A, Wang Y, Wood T, Allanore Y, Matucci-Cerinic M, Distler O, Singer O, Bush E, Fox DA, Furst DE. Abatacept in Early Diffuse Cutaneous Systemic Sclerosis: Results of a Phase II Investigator-Initiated, Multicenter, Double-Blind, Randomized, Placebo-Controlled Trial. Arthritis Rheumatol. 2020 Jan;72(1):125-136. doi: 10.1002/art.41055. Epub 2019 Dec 10. PMID 31342624
- [Background] Kreuter A, Breuckmann F, Uhle A, Brockmeyer N, Von Kobyletzki G, Freitag M, Stuecker M, Hoffmann K, Gambichler T, Altmeyer P. Low-dose UVA1 phototherapy in systemic sclerosis: effects on acrosclerosis. J Am Acad Dermatol. 2004 May;50(5):740-7. doi: 10.1016/j.jaad.2003.08.026. PMID 15097958
- [Background] Gambichler T, Schmitz L. Ultraviolet A1 Phototherapy for Fibrosing Conditions. Front Med (Lausanne). 2018 Aug 27;5:237. doi: 10.3389/fmed.2018.00237. eCollection 2018. PMID 30211165
- [Background] Skrzypek-Salamon A, Lis-Swiety A, Ranosz-Janicka I, Brzezinska-Wcislo L. Localized Scleroderma Cutaneous Assessment Tool (LoSCAT) adapted for use in adult patients: report from an initial validation study. Health Qual Life Outcomes. 2018 Sep 14;16(1):185. doi: 10.1186/s12955-018-1010-z. PMID 30217204
- [Background] Khanna D, Furst DE, Clements PJ, Allanore Y, Baron M, Czirjak L, Distler O, Foeldvari I, Kuwana M, Matucci-Cerinic M, Mayes M, Medsger T Jr, Merkel PA, Pope JE, Seibold JR, Steen V, Stevens W, Denton CP. Standardization of the modified Rodnan skin score for use in clinical trials of systemic sclerosis. J Scleroderma Relat Disord. 2017 Jan-Apr;2(1):11-18. doi: 10.5301/jsrd.5000231. PMID 28516167
- [Background] Lee SJ, Wolff D, Kitko C, Koreth J, Inamoto Y, Jagasia M, Pidala J, Olivieri A, Martin PJ, Przepiorka D, Pusic I, Dignan F, Mitchell SA, Lawitschka A, Jacobsohn D, Hall AM, Flowers ME, Schultz KR, Vogelsang G, Pavletic S. Measuring therapeutic response in chronic graft-versus-host disease. National Institutes of Health consensus development project on criteria for clinical trials in chronic graft-versus-host disease: IV. The 2014 Response Criteria Working Group report. Biol Blood Marrow Transplant. 2015 Jun;21(6):984-99. doi: 10.1016/j.bbmt.2015.02.025. Epub 2015 Mar 19. PMID 25796139
- [Background] Sandqvist G, Eklund M. Hand Mobility in Scleroderma (HAMIS) test: the reliability of a novel hand function test. Arthritis Care Res. 2000 Dec;13(6):369-74. PMID 14635312
- [Background] Steen VD, Medsger TA Jr. The value of the Health Assessment Questionnaire and special patient-generated scales to demonstrate change in systemic sclerosis patients over time. Arthritis Rheum. 1997 Nov;40(11):1984-91. doi: 10.1002/art.1780401110. PMID 9365087
- [Background] Allanore Y, Bozzi S, Terlinden A, Huscher D, Amand C, Soubrane C, Siegert E, Czirjak L, Carreira PE, Hachulla E, Zanatta E, Li M, Airo P, Mendoza FA, Rosato E, Distler O; EUSTAR Collaborators. Health Assessment Questionnaire-Disability Index (HAQ-DI) use in modelling disease progression in diffuse cutaneous systemic sclerosis: an analysis from the EUSTAR database. Arthritis Res Ther. 2020 Oct 28;22(1):257. doi: 10.1186/s13075-020-02329-2. PMID 33115544